CLINICAL TRIAL: NCT01401192
Title: A Randomized Phase II Study Comparing Pemetrexed Plus Cisplatin With Gemcitabine Plus Cisplatin According to Thymidylate Synthase Expression in Non-squamous Non-small Cell Lung Cancer
Brief Title: Pemetrexed/Cisplatin Versus Gemcitabine/Cisplatin According to Thymidylate Synthase Expression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Myung-Ju Ahn, M.D., Ph.D., Samsung medical center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-06-006
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: thymidylate synthase
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- TS positive cohort & Gem/Cis Tx arm (Experimental): Among TS expression positive patients, some will be randomized to Gem/cis therapy
  Interventions: Drug: Gemcitabine plus cisplatin
- TS+ cohort & Pem/Cis arm (Active Comparator): Among patients with TS+, randomised to Pem/cis chemotherapy
  Interventions: Drug: pemetrexed plus cisplatin
- TS negative cohort & Pem/Cis Tx arm (Active Comparator): Among patients with TS-, some will be randomised to Pem/cis Tx arm
  Interventions: Drug: pemetrexed plus cisplatin
- TS negative cohort & Gem/Cis Tx arm (Experimental): Among patients with TS-, some will be randomised to Gem/Cis Tx arm
  Interventions: Drug: Gemcitabine plus cisplatin

INTERVENTIONS:
Drug: Gemcitabine plus cisplatin — Gemcitabine 1000mg/m2 D1, D8 & cisplatin 70mg/m2 D1 every 3 weeks
  Arms: TS positive cohort & Gem/Cis Tx arm
Drug: pemetrexed plus cisplatin — Pemetrexed 500mg/m2 & cisplatin 70mg/m2 D1 every 3 weeks
  Arms: TS+ cohort & Pem/Cis arm
Drug: pemetrexed plus cisplatin — pemetrexed 500mg/m2 & cisplatin 70mg/m2 every 3 weeks
  Arms: TS negative cohort & Pem/Cis Tx arm
Drug: Gemcitabine plus cisplatin — Gemcitabine 1000mg/m2 D1, D8 & cisplatin 70mg/m2 D1 every 3 weeks
  Arms: TS negative cohort & Gem/Cis Tx arm

SUMMARY:
This study trys to evaluate the predictive role of thymidylate synthase expression for pemetrexed/cisplatin in Non-small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed nonsquamous NSCLC
* Stage IIIb, IV or recurrent NSCLC
* Age ≥ 18years
* ECOG performance status of 0 to 1
* Known TS immunohistochemical analysis data
* At least one measurable lesion by RECIST 1.1
* No previous chemotherapy or therapy with EGFR TKIs for advanced NSCLC
* Asymptomatic brain metastasis or symptomatic brain metastasis treated with local treatment such as operation, whole brain radiotherapy, or gamma-knife surgery
* At least 2 weeks later after whole brain radiotherapy or palliative radiotherapy
* Adequate renal function: estimated creatinine clearance ≥ 50mL/min

Exclusion Criteria:

* Patients whose disease recurred within 6 months after the completion of adjuvant chemotherapy.
* Patients with post-obstructive pneumonia or uncontrolled serious infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
predictive value of TS expression | 12 months
  To determine the predictive value of thymidylate synthase expression in NSCLC patients treated with pemetrexed combination therapy by interaction P value

SECONDARY OUTCOMES:
response rate | 12 months
  Whether the response rate of CG regimen is higher than that of CP regimen in TS+ patients
response rate | 12 months
  Whether the response rate of CP regimen is higher than that of CG regimen in TS- patients

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ju Ahn, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Sun JM, Ahn JS, Jung SH, Sun J, Ha SY, Han J, Park K, Ahn MJ. Pemetrexed Plus Cisplatin Versus Gemcitabine Plus Cisplatin According to Thymidylate Synthase Expression in Nonsquamous Non-Small-Cell Lung Cancer: A Biomarker-Stratified Randomized Phase II Trial. J Clin Oncol. 2015 Aug 1;33(22):2450-6. doi: 10.1200/JCO.2014.59.9324. Epub 2015 Jun 29. PMID 26124486